CLINICAL TRIAL: NCT03385109
Title: The TransEnterix European Patient Registry for Robotic Assisted Laparoscopic Procedures in Urology, Abdominal Surgery, Thoracic and Gynecologic Surgery
Brief Title: The TransEnterix European Patient Registry
Acronym: TRUST
Status: Recruiting | Type: Observational
Sponsor: Asensus Surgical (Industry)
Collaborators: RQM+ (Industry)
Responsible Party: Sponsor
Other Study IDs: TRUST
Record Dates: First submitted 2017-12-20; First posted 2017-12-28 (Actual); Last update posted 2025-09-16 (Actual); Status verified 2025-09

CONDITIONS: Surgery
Keywords: Robotic; Laparoscopic
MeSH Terms: interventions — Surgical Procedures, Operative

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 30 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- Senhance Treated: All patients enrolled who go on to have a surgery in which the Senhance system is used
  Interventions: Device: Surgery

INTERVENTIONS:
Device: Surgery — Patients are approached surgically with the Senhance Surgical System

SUMMARY:
An open label observational registry trial in which participating centers enroll subjects who had or will have a laparoscopically assisted surgery using the Senhance Surgical System.

DETAILED DESCRIPTION:
This is a prospective multi-center registry in which sites may also choose to retrospectively enroll subjects meeting the inclusion criteria, but whom have already been treated using the Senhance system. The data collection includes baseline patient characteristics, surgical details, and adverse events. Patient follow-up time point is open to the clinical practice of each center and only adverse events are tracked post discharge.

ELIGIBILITY:
Inclusion Criteria:

* patients 18-80 years old
* Signed the informed consent
* life expectancy 12 months or more

Exclusion Criteria:

-

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients at a participating center who have had or are scheduled to have surgery using the Senhance system
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2017-07-25 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2028-03 (Estimated)

PRIMARY OUTCOMES:
Adverse Event | Surgery to 30 days post op
  Any untoward sign symptom or disease

CONTACTS AND LOCATIONS:
Locations (1):
- St. Marien-Krankenhaus, Siegen, Germany

IPD SHARING:
Plan to Share IPD: No